CLINICAL TRIAL: NCT02778256
Title: Study of the Effectiveness of Vestibular Stimulation as a Coadjuvant Treatment in the Depressive Phase of Bipolar Disorder
Brief Title: Study of the Effectiveness of Vestibular Stimulation Treatment in the Depressive Phase of Bipolar Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vest Brain,Centro de Estudios Neurovestibulares (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VESTBRAIN001
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Bipolar Disorder; Depression, Bipolar
Keywords: depression, bipolar disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vestibular stimulation (Experimental): Patients of this group will receive a specific vestibular stimulation technique.
  Interventions: Device: Vestibular stimulation
- Sham vestibular stimulation (Sham Comparator): This group of patients will receive sham vestibular stimulation, similar to experimental group vestibular stimulation in the range of under threshold frequencies undistinguished from real vestibular stimulation. The absence of vestibular nystagmic response confirms that the stimulus is sham.
  Interventions: Device: Sham vestibular stimulation

INTERVENTIONS:
Device: Vestibular stimulation — A specific vestibular stimulation technique is applied to the experimental group
  Arms: Vestibular stimulation
Device: Sham vestibular stimulation — Sham vestibular stimulation using lower than threshold stimuli. The absence of vestibular nystagmus confirms that it is sham.
  Arms: Sham vestibular stimulation

SUMMARY:
Vestibular stimulation has been shown to be a very effective noninvasive treatment for major depression. Bipolar disorder is a mental illness that presents cyclic sequences of depressive and euphoric states. Depressive phases of bipolar disorder are difficult to treat and usually are resistant to actual available treatments. This study investigates the effectiveness of a particular technique of vestibular stimulation in a group of 120 bipolar type I and II patients. After randomization 60 of them will receive specific vestibular stimulation (experimental group) and 60 will receive a sham vestibular stimulation.The study will conducted in Vest Brain, Centro de Estudios Neurovestibulares, in Chile.

ELIGIBILITY:
Inclusion Criteria:

* males
* females
* 3 previous weeks with depression symptoms.
* bipolar disorder type I actual depressive phase
* bipolar disorder type II actual depressive phase
* Montgomery Asberg depression scale(MADRS) score equal or more than 20
* stable psychiatric medication during 2 weeks previous the recruitment

Exclusion Criteria:

* pregnancy
* neurologic disorder
* drugs or alcohol abuse during the 2 weeks previous the recruitment
* presence of maniac state(Young mania scale score more than 7)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2022-05 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Remission rates of depression. | 90 days

SECONDARY OUTCOMES:
Percentage of vestibular change. | 90 days
Response rates of depression | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Soza, M.D., Principal Investigator — Vest Brain,Centro de Estudios Neurovestibulares
Locations (1):
- Vest Brain, Centro de Estudios Neurovestibulares, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers by asking for the information to Dr. Ana María Soza's email: amsozaried@vestbrain.cl
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available in December 2019-March 2020 and can be asked to Dr. Ana María Soza´s email amsozaried@vestbrain.cl
Access Criteria: The criteria to access is asking for the information to Dr. Ana María Soza´s email amsozaried@vestbrain.cl
URL: https://www.vestbrain.cl